CLINICAL TRIAL: NCT02144740
Title: A Study of Two Parts to Determine the Effect of NWT-03 on Blood Pressure in Healthy Subjects
Brief Title: Effect of NWT-03 on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newtricious R&D BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AFCRO-041 - Part 2
Record Dates: First submitted 2013-11-06; First posted 2014-05-22 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Blood Pressure; Albuminuria
Keywords: Flow-mediated dilation
MeSH Terms: conditions — Albuminuria | interventions — NWT-03

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NWT-03, then placebo (Other): 4 weeks 2g NWT-03 followed by placebo , separated by a 4wk wash-out period
  Interventions: Dietary Supplement: NWT-03, an egg-white protein hydrolysate; Dietary Supplement: Placebo
- Placebo, then NWT-03 (Other): 4 weeks placebo followed by 2g NWT-03, separated by a 4wk wash-out period
  Interventions: Dietary Supplement: NWT-03, an egg-white protein hydrolysate; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NWT-03, an egg-white protein hydrolysate — For placebo comparator, a combination of sweetener + aroma, which was equal to the combination used in the intervention period, was given
Dietary Supplement: Placebo — A combination of sweetener + aroma , which was equal to the combination used in the intervention period, was given.

SUMMARY:
Part 2 of the study will assess the effect of 2g of NWT-03 (an egg-white protein hydrolysate) on systolic and diastolic blood pressure and flow-mediated dilation in a crossover designed study in healthy adults with mild hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent,
* Be between 35 and 75 years of age,
* Be in generally good health as determined by the investigator,
* Smokers and non-smokers are eligible,
* Have a stable body weight (< 5% change) over the past 3-months,
* Have a Body Mass Index (BMI) between 25 and 35 kg/m2,
* Be mild hypertensive (Systolic Blood Pressure 140-159 mmHg & Diastolic Blood Pressure 80-99 mmHg).

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the below criteria;

1. Are less than 35 and greater than 75 years of age,
2. Females are pregnant, lactating or wish to become pregnant during the study. Female subject is currently either of:

   1. non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or any female who is surgically sterilized (via documented hysterectomy or bilateral tubal ligation). (For purposes of this study, postmenopausal is defined as one year without menses), OR
   2. child bearing potential, the subject is eligible to enter and participate in this study if she is not lactating and has a negative urine pregnancy test at the screening visit, visit 2 and upon completion of the study at visit 7. The subject must also agree to one of the following methods of contraception:

      * Complete abstinence from intercourse two weeks prior to administration of study drug, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the study medication in cases where subject discontinues the study prematurely. (Subjects utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit.) or,
      * has a male sexual partner who is surgically sterilized prior to the Screen Visit and is the only male sexual partner for that subject or,
      * sexual partner(s) is/are exclusively female or,
      * Oral contraceptives (either combined or progestogen only) with double-barrier method of contraception consisting of spermicide with either condom or diaphragm. (Women of child-bearing potential using an oral contraceptive in combination with a double-barrier method of contraception are required to continue to use this form of contraception for 1 week following discontinuation of study medication).
      * Use of double-barrier contraception, specifically, a spermicide plus a mechanical barrier (e.g. male condom, female diaphragm). The subject must be using this method for at least 1 week following the end of the study or,
      * Use of any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year. The subject must have the device inserted at least 2 weeks prior to the first Screen Visit, throughout the study, and 2 weeks following the end of the study.
3. Are hypersensitive to any of the components of the test product,
4. Have a significant acute or chronic coexisting illness such as cardiovascular disease, Chronic kidney disease (CKD), gastrointestinal disorder, endocrinological disorder, immunological disorder, metabolic disease or any condition which contraindicates, in the investigators judgement, entry to the study,
5. Having a condition or have taken a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; to include diuretics, blood pressure medication and medication interfering with renin-angiotensin-aldosterone system (RAAS), such as ACE-inhibitors, angiotensin receptor blockers, direct renin inhibitors or aldosterone receptor inhibitor,
6. Are taking non-steroidal anti-inflammatory drugs (NSAIDs) within 2 weeks of baseline visit or for the duration of the trial,
7. Suffer from diabetes mellitus, either type I and type II,
8. Consume more than the recommended alcohol guidelines i.e. >21 alcohol units/week for males and >14 units/week for females,
9. History of illicit drug use,
10. Use of nasal decongestants and other over-the counter or herbal preparation within 2 weeks of baseline visit and for the duration of the trial,
11. Heavy intake of coffee (i.e. more than 4 cups daily) within 2 weeks of baseline visit and for the duration of the trial,
12. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial,
13. Subjects may not be receiving treatment involving experimental drugs,
14. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study. An exception will be made where subjects have participated in part 1 of the study,
15. Have a malignant disease or any concomitant end-stage organ disease.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in daytime systolic blood pressure at 4 and 8 weeks | For both intervention periods: 48h ABPM before baseline visit, 4 and 8 weeks after baseline visit

SECONDARY OUTCOMES:
Change from baseline in daytime diastolic blood pressure at 4 and 8 weeks | For both intervention periods: 48h ABPM before baseline visit, 4 and 8 weeks after baseline visit
Change from baseline in flow-mediated dilation (only for n=10 subgroup) at 8 weeks | Both periods: at baseline and after 8 weeks
Change from 48 before baseline in albuminuria at 8 weeks | For each period: 48h before baseline and 8 weeks after baseline

OTHER OUTCOMES:
Vitals (weight, height, BMI) | During screening (up to 4 weeks before baseline)
eGFR | Each period: 48h before baseline and week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Food CRO, Cork, Ireland